CLINICAL TRIAL: NCT06942806
Title: The Efficacy of High-frequency Short-time Spinal Cord Stimulation in the Treatment of Herpes Zoster-associated Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Li Zhao (Other)
Responsible Party: Sponsor-Investigator, Li Zhao, Attending Physician, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Other Study IDs: 20241212
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Herpes Zoster Pain
Keywords: Spinal cord stimulation; Herpes zoster-associated neuralgia; Neuromodulation; High-frequency spinal cord electrical stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF group: HF-SCS parameter settings: Frequency 1000 Hz, pulse width 60-180 μs, amplitude 0.5-3.0 V
  Interventions: Other: HF-SCS parameter settings: Frequency 1000 Hz, pulse width 60-180 μs, amplitude 0.5-3.0 V
- LF group: LH-SCS parameter settings: Frequency 30-100 Hz, pulse width 100-300 μs, amplitude 0.5-5.0 V
  Interventions: Other: LH-SCS parameter settings: Frequency 30-100 Hz, pulse width 100-300 μs, amplitude 0.5-5.0 V

INTERVENTIONS:
Other: HF-SCS parameter settings: Frequency 1000 Hz, pulse width 60-180 μs, amplitude 0.5-3.0 V — HF-SCS parameter settings: Frequency 1000 Hz, pulse width 60-180 μs, amplitude 0.5-3.0 V
  Groups: HF group
Other: LH-SCS parameter settings: Frequency 30-100 Hz, pulse width 100-300 μs, amplitude 0.5-5.0 V — LH-SCS parameter settings: Frequency 30-100 Hz, pulse width 100-300 μs, amplitude 0.5-5.0 V
  Groups: LF group

SUMMARY:
Zoster-associated neuralgia (ZAN) is a type of neuropathic pain caused by the reactivation of the varicella-zoster virus (VZV). The global annual incidence is approximately 3-5 per 1,000 individuals, and in China, the incidence is around 4.89 per 1,000 individuals, increasing with age. The underlying mechanisms of ZAN involve neuroinflammation, peripheral and central sensitization, and other factors, ultimately leading to anxiety, depression, and significant reductions in quality of life. Treating ZAN remains challenging.

Spinal cord stimulation (SCS) alleviates pain via multiple mechanisms, including the gate control theory, modulation of neurotransmitters (e.g., gamma-aminobutyric acid), suppression of neuroinflammation (e.g., reduced levels of IL-1β and TNF-α), and promotion of autophagy. However, traditional low-frequency SCS (30-100 Hz) is limited by incomplete pain coverage, reduced long-term efficacy, and side effects such as paresthesia (e.g., tingling sensations).

High-frequency SCS (HF-SCS, 1,000 Hz) offers pain relief without inducing paresthesia. Studies have suggested that it may be superior to traditional SCS. However, clinical data on the use of HF-SCS in ZAN are limited, and no such studies have been conducted in China.

This study aims to compare the efficacy of short-term high-frequency (1 kHz) SCS with traditional low-frequency SCS in the treatment of ZAN. By evaluating outcomes such as pain relief (NRS scores), improvements in anxiety and depression (HADS), sleep quality (PSQI), patient-reported experience, and complication rates, this research seeks to assess the safety and efficacy of short-term HF-SCS, thereby potentially providing a novel therapeutic strategy for patients with ZAN.

DETAILED DESCRIPTION:
Zoster-associated neuralgia (ZAN) refers to neuropathic pain resulting from herpes zoster (HZ) infection. Based on the duration of symptoms, ZAN is classified into three stages: acute herpetic neuralgia (AHN, less than 1 month), subacute herpetic neuralgia (SHN, 1 to 3 months), and postherpetic neuralgia (PHN, more than 3 months).The global annual incidence of HZ is approximately 3 to 5 per 1,000 individuals, with higher rates observed among individuals aged 50 years and older, and among females. In China, the annual incidence is approximately 4.89 per 1,000 individuals, with a notable increase observed with advancing age.

Pain is the most common clinical symptom of HZ, and its severity correlates with age, immune status, and initial pain intensity. Older adults and immunocompromised patients are more prone to developing PHN . HZ may also lead to complications such as ocular herpes zoster, meningitis, and motor nerve damage, particularly in immunocompromised individuals, where the risk and severity of these complications are significantly elevated . The pathogenesis of PHN remains incompletely understood and may involve inflammatory responses, ion channel alterations, and peripheral/central sensitization . Chronic pain severely impacts patients' quality of life and can lead to psychological issues such as anxiety, depression, and sleep disturbances, imposing substantial burdens on families and society .

ZAN is challenging to treat, with current approaches including pharmacotherapy, nerve blocks, pulsed radiofrequency, and spinal cord stimulation (SCS) . SCS is a minimally invasive neuromodulation technique widely used for chronic pain. It involves implanting electrodes in the epidural space to deliver electrical pulses to the dorsal columns and dorsal horn structures, thereby modulating pain signal transmission. Although the analgesic mechanism of SCS is not fully elucidated, its theoretical basis dates back to the 1965 "gate control theory" proposed by Melzack and Wall. This theory posits that activating large-diameter Aβ afferent fibers inhibits nociceptive signals mediated by small-diameter Aδ and C fibers, reducing spinal sensitization .

Recent studies suggest that SCS also regulates neurotransmitters, suppresses neuroinflammation, and modulates autophagy . At the neurotransmitter level, SCS enhances the release of γ-aminobutyric acid (GABA), reduces glutamate concentrations, amplifies endogenous opioid signaling, and activates the endocannabinoid system, thereby rebalancing dorsal horn activity and inhibiting pain transmission. In neuroinflammatory regulation, SCS elevates anti-inflammatory resolvin D1, reduces pro-inflammatory cytokines (IL-1β, TNF-α), suppresses microglial overactivation, and modulates the p38MAPK pathway, thereby attenuating neuroinflammation and pain hypersensitivity . Additionally, SCS promotes neuronal autophagy, accelerating the clearance of damaged cellular components to restore function and mitigate neural injury, further alleviating pain . These mechanisms collectively support SCS as a multimodal analgesic strategy, driving its clinical adoption.

SCS has shown efficacy in ZAN treatment, particularly for patients refractory to medications or other minimally invasive therapies. However, traditional low-frequency SCS (30-100 Hz), which relies on high-intensity pulses to modulate spinal and ascending pain pathways, often induces paresthesia (e.g., tingling) as a side effect. Clinical limitations include incomplete pain coverage, diminishing efficacy over time, and discomfort in non-target areas, necessitating novel SCS paradigms with improved efficacy and tolerability .

High-frequency spinal cord stimulation (HF-SCS) is an emerging neuromodulation technique that alleviates chronic neuropathic pain without paresthesia and may benefit patients unresponsive to traditional SCS. In China, HF-SCS research remains exploratory, with no clinical studies on ZAN. International studies, though advanced, lack systematic data on ZAN, with heterogeneous parameters (indications, frequency, pulse width, etc.). This study compares short-term 1 kHz HF-SCS with traditional low-frequency SCS in ZAN treatment, evaluating pain relief, psychological status (anxiety/depression), sleep quality, patient experience, and complication rates. The findings aim to establish the safety and efficacy of short-term HF-SCS for ZAN, offering a novel therapeutic option for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with inadequate response to non-surgical treatments such as pharmacotherapy;
2. Patients with major organ dysfunction intolerant to drug therapy;
3. Patients with systemic comorbidities (e.g., hypertension, diabetes mellitus);
4. Patients with moderate to severe pain intensity (Numerical Rating Scale [NRS] score ≥ 4).

Exclusion Criteria:

1. Patients with severe psychiatric disorders;
2. Patients with severe local or systemic infections at the puncture site;
3. Patients with severe coagulopathies (platelet count < 80×10⁹/L during puncture) or those requiring uninterrupted anticoagulation therapy without bridging protocol;
4. Patients with end-stage organ failure who cannot maintain prone positioning or tolerate the procedure;
5. Patients with severe spinal stenosis, vertebral ankylosis, or scoliosis;
6. Patients with language barrier or impaired communication abilities.ion

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with herpes zoster-associated neuralgia undergoing spinal cord electrical stimulation (SCS) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Numerical scale pain score | Preoperative, postoperative day 7, postoperative day 30, postoperative day 90, postoperative day 180.
  An NRS score of 0 indicates no pain; scores ≥1 and <4 indicate mild pain; scores ≥4 and <6 indicate moderate pain; scores ≥7 indicate severe pain.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | Preoperative, postoperative day 7, postoperative day 30, postoperative day 90, postoperative day 180.
  A 5-point Likert scale ranging from 0 to 4 is used. A total score ≥29 may indicate severe anxiety; ≥21 indicates definite marked anxiety; ≥14 indicates definite anxiety; a score above 7 may suggest anxiety; a score below 7 indicates no symptoms of anxiety.
Hamilton Depression Rating Scale | Preoperative, postoperative day 7, postoperative day 30, postoperative day 90, postoperative day 180.
  A total HAMD score of less than 7 indicates no depression; a score of 7-17 indicates mild depression; a score of 18-24 indicates moderate depression; and a score above 24 indicates severe depression.
Pittsburgh sleep quality index | Preoperative, postoperative day 7, postoperative day 30, postoperative day 90, postoperative day 180.
  The total PSQI score ranges from 0 to 20, with lower scores indicating better sleep quality. It is used to assess overall sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- 149 Dalian Road, Huichuan District, Zunyi City, Guizhou Province, Zunyi, Guizhou, China